CLINICAL TRIAL: NCT03358940
Title: Assessment of Non-medical Use of Misoprostol in Case of Miscarriage or Threatened Miscarriage in Guadeloupe.
Brief Title: Assessment of Non-medical Use of Misoprostol in Case of Miscarriage or Threatened Miscarriage.
Acronym: MISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBM-PAP-2015/31
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Threatened Miscarriage
Keywords: Non-medical abortion; Misoprostol; miscarriage complications; Guadeloupe
MeSH Terms: conditions — Abortion, Threatened | interventions — Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: Will be included in the student a patient who is maximum 24 weeks pregnant with miscarriage complications or not, or threatened miscarriage, or voluntary termination of pregnancy using misoprostol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with miscarriage complications or not (Other): The day of inclusion, for patient with miscarriage complications or not, or threatened miscarriage there will be a urine collection. In case of hospitalization, another urine collection will be done between 12 and 18 hours after the inclusion. For patient coming for voluntary termination of pregnancy using misoprostol, a urine collection will be done the day of the inclusion and another ones 1, 4, 12 and 24 hours after the inclusion.
  Interventions: Other: urine collection

INTERVENTIONS:
Other: urine collection — For patient with miscarriage complications or not, or threatened miscarriage there will be a urine collection the day of the inclusion. In case of hospitalization, another urine collection will be done between 12 and 18 hours after the inclusion. For patient coming for voluntary termination of pregnancy using misoprostol, a urine collection will be done the day of the inclusion and another ones 1, 4, 12 and 24 hours after the inclusion.

SUMMARY:
Non-medical used of misoprostol for abortion is a growing concern in Guadeloupe. Such situation is reasonable for countries in which abortion is not easy to obtain or prohibited. However regarding the risk of complications, it is less understandable in region like Guadeloupe where legal abortion with medical assistance is accessible for all and free.

The aim of the study is to investigate on the amount of misoprostol taken by women in Guadeloupe, by doing an analytical measurement. The aim is to evaluate batter this practice in Guadeloupe, when the main objective of the study is to detect the presence or the absence of misoprostol in the urine sample of the woman coming at hospital for threatened miscarriage or miscarriage complications. Moreover, these abortions can be more important than spontaneous miscarriage.

DETAILED DESCRIPTION:
Previous assessments in many countries as well in Guadeloupe were based on self-declaration. Such assessment is suspected to lead to underestimation. In addition, to our knowledge, no comparison has been done between those induced abortions and the natural miscarriages.

Illegal aspects of non-medical use of misoprostol and consequently bad self-declaration are hindrance to good assessment of the burden of such practice among patients asking for medical care at emergency unit for miscarriage or threatened miscarriage. They may also impair quality of evaluation of the relative risk associated to miscarriage threatened miscarriage induced by misoprostol compared to the same obstetrical complication without absorption of misoprostol. After a dose, misoprostol is quickly active and metabolised. It is mainly eliminated in urine. This elimination seems to be a way to increase the length of detection of the use of misoprostol. The aim of our study is to perform a detection of misoprostol in urine sample of patients hospitalised for a miscarriage or threatened miscarriage. This sample will be done during emergency cares. The study will not change the procedure of medical care of the patients during or after hospitalisation. All data will be obtained from information and result of tests normally done in such situation.

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria:
* All patients who come at the maternity emergency unit for miscarriage or threatened miscarriage by 24 weeks of amenorrhea or patient receiving misoprostol for voluntary abortion.
* Age ≥ 12 years old
* Patient insured under the French social security system

Exclusion Criteria:

* Refusal to participate in the study
* Age < 12 years old

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only pregnant women can be included in the study.
Enrollment: 210 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Detection of misoprostol in urine sample | Enrollment visit
  A descriptive analysis of variable is planned. And comparison between exposed or non-exposed to misoprostol will be done. Uni and multivariate linear regression will be used for analyse associated risk of misoprostol use.

SECONDARY OUTCOMES:
sociodemographic feature of patient and medical outcomes of the miscarriage or threatened miscarriage. | Enrollment visit
  A descriptive analysis of variable is planned. And comparison between exposed or non-exposed to misoprostol will be done. Uni and multivariate linear regression will be used for analyse associated risk of misoprostol use.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe KADHEL, medicine degree, gynecology, Principal Investigator — Hospital University Center of Pointe-à-Pitre

IPD SHARING:
Plan to Share IPD: No